CLINICAL TRIAL: NCT00706823
Title: A Randomized Clinical Comparison of the Intersurgical I-gel and the Laryngeal Mask Airway Unique in Non-Obese Adult Patients During General Surgery
Brief Title: Comparison of I-gel to the Laryngeal Mask Airway
Acronym: I-gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Carin A. Hagberg, ◦Professor and Chairman, Joseph C. Gable, MD Endowed Chair, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-08-0004
Record Dates: First submitted 2008-06-24; First posted 2008-06-30 (Estimated); Results first posted 2011-04-05 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-01

CONDITIONS: Endotracheal Intubation; Supraglottic Airway
Keywords: Endotracheal Intubation; Supraglottic Airway

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- i-gel-SGA (Experimental): Patients who received i-gel supraglottic device (i-gel airway) for intubation
  Interventions: Device: i-gel airway (Intersurgical Ltd., Wokingham, England)
- LMA-Unique (Active Comparator): Patients who received the Laryngeal Mask Airway-Unique (uLMA) for intubation
  Interventions: Device: Laryngeal Mask Airway-Unique

INTERVENTIONS:
Device: i-gel airway (Intersurgical Ltd., Wokingham, England) — supra-glottic airway device
  Arms: i-gel-SGA
Device: Laryngeal Mask Airway-Unique — supra-glottic airway device
  Arms: LMA-Unique

SUMMARY:
The purpose of this study is to evaluate a new disposable supra-glottic airway device, the i-gel airway (Intersurgical Ltd., Wokingham, England). We propose to test its ease of insertion, position within the airway, drain tube patency and anatomic sealing properties during mechanical ventilation in non-obese anesthetized patients undergoing elective general surgery. The study device will be compared to the current standard in the industry, the LMA Unique.

DETAILED DESCRIPTION:
During the past decade, several pharyngeal airways have been introduced for airway management, such as the Laryngeal Mask Airway (LMA), the Cobra perilaryngeal airway, the Esophageal Tracheal Combitube (ETC), the EasyTube, the Laryngeal Tube6, and the Streamlined Liner of the Pharyngeal Airway (SLIPA). These airway devices have become very popular because of their ability to maintain an airway without perturbing the trachea and can be used in patients without muscle relaxation who are only lightly anesthetized.

The LMA Classic (cLMA) generally provides an adequate airway, but certain problems remain:

1. In 8-33% of LMA placements, more than one attempt is required.
2. It is sometimes difficult to advance the LMA without extending the neck (which is contraindicated in some patients).
3. The device does not protect the airway from aspiration of gastric contents.
4. It does not provide an airtight seal around the larynx (the usual pressures causing leakage of gas being 15-20 cm H20). Consequently, the device may function poorly during positive-pressure ventilation.
5. The esophagus is included within the rim of the LMA in 10-15% of patients, directly exposing the esophagus to positive airway pressures. This often results in insufflation of the stomach and postoperative discomfort.

The LMA Unique (uLMA) is a disposable, inflatable supraglottic airway device that is based on the LMA Classic design which has been used as the "model" in the industry. It has been listed as a commonly accepted device for routine and rescue airway management and is now listed in the American Society of Anesthesiologists (ASA) Difficult Airway Management Algorithm as an airway conduit for tracheal intubation.

The i-gel (Intersurgical Ltd., Wokingham, England) is a cuffless, single-use supraglottic airway device designed to provide a more effective seal than the uLMA, thus eliminating problems 3-5 described above with the addition of a gastric drain. Made of a gel-like thermoplastic elastomer, the i-gel has an anatomically-designed mask that allows quick, easy insertion and can accurately position itself over the laryngeal framework to provide a reliable perilaryngeal seal without the need for an inflatable cuff. In a preliminary study, the peak airway pressures were found to be above 30 cm H2O with a sustained leak pressure of 24 cm H2O versus an average of 18-21 cm H2O seen with the cLMA. According to the 100 patient trial, the i-gel is easier to insert, it has better sealing properties and there is no cuffed inflates.

This clinical study has been designed to compare the i-gel and the uLMA, as to ease of placement, ventilation during mechanical ventilation, proper positioning, seal pressures, the patency of the drain tube, and finally, any complications with their use. Fiberoptic observations through each device will provide information in relation to the epiglottis and the distal opening of the device.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects will be adult surgical candidates aged 18-80, ASA I-II, Mallampati I or II, presenting for elective surgery who require general anesthesia in whom tracheal intubation is not necessary.
2. Both male and female patients will be included.

Exclusion Criteria:

Patients will be excluded from the study if they present as Mallampati III or IV, ASA III-V or emergency status. Additionally, they will be excluded if they meet one of the contraindication criteria of the LMA including:

1. obesity, (BMI > 35 kg/m2)
2. pregnancy
3. history of gastric regurgitation, heart burn, ileus or "full stomach"
4. history of low pulmonary compliance or high pulmonary resistance
5. known history of difficult endotracheal intubation or signs suggesting the possibility of difficult intubation
6. pharyngeal pathology
7. upper airway obstruction due to laryngeal pathology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carin A Hagberg, M.D., Principal Investigator — The University of Texas Medical School at Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients for this study have been recruited from Feb 2008 through July 2008. The patients were recruited from the day surgery and holding areas.
Groups:
- I-gel-SGA: Patients who received i-gel for intubation. The i-gel is a disposable, cuffless, single-use supraglottic airway device used for airway management. It is similar to the uLMA with the addition of a gastric drain. The i-gel is made of a gel-like thermoplastic elastomer, has an anatomically-designed mask that allows quick and easy insertion, and can accurately position itself over the laryngeal framework to provide a reliable perilaryngeal seal without the need for an inflatable cuff.
- LMA-Unique: Patients who received LMA Unique (uLMA) for intubation. The uLMA is a disposable, inflatable supraglottic airway device that is based on the LMA Classic design, which has been used as the "model" in the industry. It has been listed as a commonly accepted device for routine and rescue airway management and is now listed in the American Society of Anesthesiologists (ASA) Difficult Airway Management Algorithm as an airway conduit for tracheal intubation.
Period: Overall Study
Arm/Group | I-gel-SGA | LMA-Unique
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- I-gel-SGA: Patients who received i-gel SGA for intubation
- LMA-Unique: Patients who received LMA-Unique for intubation
- Total: Total of all reporting groups
Arm/Group | I-gel-SGA | LMA-Unique | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 25 | 23 | 48
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (10.5) | 35.3 (16.6) | 37.28 (13.8)
Gender [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 16 | 19 | 35
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Time Required for Intubation
Description: The total time to intubation was measured from the beginning of supraglottic airway device (SGA) insertion to successful endotracheal tube intubation, verified by detection of CO2 on the capnogram (anesthesia machine).
Time Frame: duration of intubation
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | I-gel-SGA | LMA-Unique
Number analyzed (Participants) | 25 | 25
seconds | 21.04 (12.6) | 30.04 (14.1)
Statistical Analysis 1: Comparison: I-gel-SGA vs LMA-Unique; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

2. Secondary Outcome: Level of Difficulty for Intubation
Description: Ease of SGA insertion and intubation was subjectively assessed by the operator on a scale from 1 to 5 (1 = very easy, 2 = easy, 3 = neutral, 4 = difficult, 5 = very difficult).
Time Frame: duration of intubation
Measure: Number; unit: participants
Arm/Group | I-gel-SGA | LMA-Unique
Number analyzed (Participants) | 25 | 25
participants
  Very Easy | 11 | 8
  Easy | 12 | 17
  Neutral | 0 | 0
  Difficult | 2 | 0
  Very Difficult | 0 | 0
Statistical Analysis 1: Comparison: I-gel-SGA vs LMA-Unique; Test type: Superiority or Other; p = 0.22, Fisher Exact

3. Secondary Outcome: Number of Participants With Oropharyngeal Discomfort
Description: Oropharyngeal discomfort was assessed. including sore throat, hoarseness, and dysphagia.
Time Frame: post operative, immediately and 24 hrs after intubation
Measure: Number; unit: participants
Arm/Group | I-gel-SGA | LMA-Unique
Number analyzed (Participants) | 25 | 25
participants
  Postop symptoms present | 6 | 10
  Postop symptoms absent | 19 | 15

4. Primary Outcome: Leak Pressure
Description: After successful placement, airway leak pressure was assessed by closing the circuit to atmosphere and allowing fresh gas flow to build airway pressure. The pressure at which an audible leak was heard was recorded; airway pressure was not permitted to exceed 40 cm H2O.
Time Frame: duration of intubation
Measure: Mean (Standard Deviation); unit: cm of H2O
Arm/Group | I-gel-SGA | LMA-Unique
Number analyzed (Participants) | 25 | 25
cm of H2O | 23.08 (7.3) | 20.88 (4.5)
Statistical Analysis 1: Comparison: I-gel-SGA vs LMA-Unique; Test type: Superiority or Other; p = 0.22, t-test, 2 sided

5. Secondary Outcome: Number of Participants With Successful Gastric Drainage Tube Placement as Assessed by Fiberoptic Scope Visualization
Description: When the fiberoptic scope was placed in the gastirc drain tube of the i-gel, if the esophageal mucosa was visible and the stomach was readily accessible, then placement was considered succussful.
Time Frame: after intubation
Population: Only the -gel has a gastric drainage tube--the uLMA does not. Thus, only those receiving the i-gel were assessed for this measure.
Measure: Number; unit: participants
Arm/Group | I-gel-SGA | LMA-Unique
Number analyzed (Participants) | 25 | 0
participants
  Esophageal mucosa visible and stomach accessible | 22 |
  Upper esophageal sphincter visible | 2 |
  Glottis visible | 1 |

6. Secondary Outcome: Number of Attempts
Description: The number of attempts taken to place the device
Time Frame: Before intubation
Measure: Number; unit: participants
Arm/Group | I-gel-SGA | LMA-Unique
Number analyzed (Participants) | 25 | 25
participants
  1 attempt | 17 | 21
  2 attempts | 7 | 3
  3 attempts | 1 | 1
Statistical Analysis 1: Comparison: I-gel-SGA vs LMA-Unique; Test type: Superiority or Other; p = 0.03, Regression, Logistic; Odds Ratio (OR) = 8.11, 95% CI 2-sided [1.1 to 58.6]

ADVERSE EVENTS:
Time Frame: Postoperatively, within 2 hours of emergence and extubation
Arm/Group | I-gel-SGA | LMA-Unique
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 6/25 | 10/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | I-gel-SGA (N=25) | LMA-Unique (N=25)
Oropharyngeal discomfort (Surgical and medical procedures) | 6 (25) | 10 (25) — Oropharyngeal discomfort, including sore throat, hoarseness, and dysphagia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No